CLINICAL TRIAL: NCT07178457
Title: Brentuximab Vedotin in CutAneous T-cell Lymphomas (CTCL): Post-allogeneic Hematopoietic Stem Cell Transplant Maintenance
Acronym: BeCALM
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APHP241010
Record Dates: First submitted 2025-08-25; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Cutaneous T Cell Lymphoma (CTCL); Brentuximab Vedotin
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous | interventions — Brentuximab Vedotin

STUDY DESIGN:
Intervention Model Description: Multicentre, prospective, double-blind, placebo-controlled, (ratio 1:1) randomized study, with randomization stratified on donor type, previous use of BV or not and Complete Response (CR)/Partial Response (PR)/Stable disease (SD) after 1st course of BV
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brentuximab vedotin (Experimental)
  Interventions: Drug: Brentuximab Vedotin (Bv)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Brentuximab Vedotin (Bv) — 1.8 mg/kg in 100 mlof NaCl 0.9%, Q3W with a maximum of 16 cycles
  Arms: Brentuximab vedotin
Drug: Placebo — NaCl 0.9% 100 ml IV Q3W with a maximum of 16 cycles
  Arms: Placebo

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (alloHSCT) showed efficacy in advanced-stage, high-risk, treatment sensitive cutaneous T-cell lymphomas (CTCL) in a prospective, propensity score-matched controlled study (CUTALLO) published by our group in the Lancet in 2023. Nevertheless, it is associated with a high rate of early relapse, with 2-year progression-free survival around 30%. Brentuximab vedotin (BV) has shown efficacy in the treatment of CD30-expressing CTCL after at least one prior systemic treatment in the ALCANZA trial and is market approved in this indication in Europe and the United States of America. BV has been successfully used as salvage treatment in the post-transplant setting in advanced CTCL. It has been shown that 90% of CTCL express CD30. To reduce the incidence of post-allograft relapse, we propose to assess the routine use of BV post-allograft in adult patients with advanced CD30-expressing mycosis fungoides-CTCL, who have received at least one line of prior systemic therapy, compared to placebo. Switch will be allowed from placebo to BV in case of disease progression. This project is supported by well-organized research networks with a strong track-record of published results in the field: French Study Group on Cutaneous Lymphomas (GFELC, Groupe Français d'Etude des Lymphomes Cutanés), INCa-labelled national rare cancers network; and the French Society of Bone Marrow Transplantation and CellTherapy. In the post-transplant setting, the current state-of-the-art practice is to treat patients once they have relapsed post-allogeneic transplant, whereas no prophylactic treatment is given at the time in the absence of characterized disease relapse. This ethically and scientifically justifies the proposal to evaluate whether earlier, prophylactic treatment with BV increases progression-free survival compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for study entry, patients must meet all of the following criteria:

* Age ≥ 18 and ≤ 70 years
* Histopathologically confirmed diagnosis of ISCL-EORTC stage IIB, III, IVA or IVB MF (mycosis fungoides) with ≥1% CD30 expression determined by immunohistochemistry
* ECOG performance status 0-1
* Relapsed or refractory to at least one line of systemic treatment
* Complete or partial response of the lymphoma at the time of study inclusion
* Having received recent alloHSCT from a sibling, 10/10 or 9/10 phenoidentical, or haploidentical donor (60 to 90 days before inclusion)
* Adequate liver function:

  * Total bilirubin ≤ 2 xULN, or Direct bilirubin ≤ 2xULN if total bilirubin is >2xULN, or total bilirubin >2 xULN if elevated total bilirubin is attributed to Gilbert's syndrome
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x ULN
* Adequate hematological function:

  * Absolute neutrophil count of ≥ 1.0 G/L
  * Platelet count of ≥ 50 G/L
  * Hemoglobin ≥ 9 g/dL
* Adequate renal function: creatinine clearance calculated by Cockcroft & Gault formula of ≥ 50 mL/min
* Patient affiliated to life insurance
* Written informed consent given by the patient

Exclusion Criteria:

Any of the following criteria requires the exclusion of the patient before randomization:

* Second or higher allogeneic HSCT,
* Other progressive neoplastic or psychotic disease,
* Left ventricular ejection fraction < 50%, carbone monoxide diffusion capacity < 50% of the theoretical value,
* History of BV-induced adverse event without resolution to current grade <2. Previous treatment with brentuximab vedotin alone, in the absence of current ≥ grade 2 BV-induced side effect, is NOT an exclusion criterion.
* History of disease refractoriness, progression or relapse during BV treatment. Previous treatment with BV alone, if the disease was treatment-sensitive (complete, partial response or stable disease), is NOT an exclusion criterion.
* History of ≥ grade 4 adverse event induced by BV. Previous <grade 4 adverse event induced by BV is not an exclusion criterion if the adverse event has regressed to grade<2.
* Contra-indication to BV including current >grade 2 neutropenia or active infection,
* Progressive disease or relapse at study inclusion compared to the screening visit status,
* Refusal of highly effective birth control method for female participant of childbearing potential and male participant with a female partner of childbearing potential,
* Pregnant and/or breastfeeding women,
* Participation to another interventional clinical trial,
* Adults subject to a legal protection measure (guardianship, curatorship and safeguard of justice),
* Patients deprived of their liberty by a judicial or administrative decision

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2032-11-01 (Estimated); Study Completion 2032-11-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 2 years after randomization

SECONDARY OUTCOMES:
Overall survival | 2 years after randomization
Quality of life scoring | At 1 year
  The EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30) is a 30-item scale with scores ranging from 0 to 100. A higher score indicates better quality of life.
Quality of life scoring | At 1 year
  The Skindex-29 is a 29-item questionnaire assessing the impact of skin diseases on quality of life, with scores ranging from 0 to 100. Higher scores indicate greater impairment in quality of life.
Cumulative incidence of disease relapse | At 2 years
Cumulative incidence of acute graft-versus-host disease (GVHD) | At 2 years
Cumulative incidence of chronic GVHD | At 2 years
Cumulative incidence of non-relapse mortality | At 2 years
Quality of life scoring | At 2 years
  The EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30) is a 30-item scale with scores ranging from 0 to 100. A higher score indicates better quality of life.
Quality of life scoring | At 2 years
  The Skindex-29 is a 29-item questionnaire assessing the impact of skin diseases on quality of life, with scores ranging from 0 to 100. Higher scores indicate greater impairment in quality of life.

IPD SHARING:
Plan to Share IPD: Undecided